CLINICAL TRIAL: NCT06582264
Title: A Phase 1b, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate Safety, Engraftment, and Initial Signs of Clinical Activity of MB310 in Patients With Active, Mild-to-Moderate Ulcerative Colitis
Brief Title: A Phase 1b Trial to Evaluate the Safety of MB310 in Patients With Active, Mild-to-Moderate Ulcerative Colitis
Acronym: COMPOSER-1
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Microbiotica Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB310-01; 2023-507376-50 (EudraCT Number)
Record Dates: First submitted 2024-08-19; First posted 2024-09-03 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vancomycin preconditioning followed by MB310 (Experimental): Vancomycin 125mg QID for 5 days plus 2 day wash-out prior to receiving MB310 PO (2 capsules once a day) for 12 weeks
  Interventions: Biological: MB310; Drug: Vancomycin
- Vancomycin preconditioning followed by Placebo (Placebo Comparator): Vancomycin 125mg QID for 5 days plus 2 day wash-out prior to receiving MB310-matching placebo PO (2 capsules once a day) for 12 weeks
  Interventions: Other: Placebo; Drug: Vancomycin

INTERVENTIONS:
Biological: MB310 — Live bacterial therapeutic for oral administration
  Arms: Vancomycin preconditioning followed by MB310
Other: Placebo — MB310-matching placebo for oral administration
  Arms: Vancomycin preconditioning followed by Placebo
Drug: Vancomycin — Antibiotic

SUMMARY:
A Phase 1b study to evaluate the safety and tolerability of MB310 given to patients who have active mild-to-moderate ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Must be aged 18 to 70 years, inclusive, at the time of signing informed consent;
* Must have newly diagnosed or a history of recurrent UC based on clinical, endoscopic, and histological assessments;
* Must have active, mild-to-moderate UC as defined by the Modified Mayo Score (MMS) of ≥4 and ≤7, and an Endoscopic Subscore of ≤2 in the most affected area proximally ≥15 cm from anal verge;
* Male patients, and female patients of childbearing potential who are at risk of pregnancy, must agree to use a highly effective method of birth control
* Female patients must not be pregnant or breastfeeding;
* Male patients must agree to abstain from sperm donation;
* Must be able to understand and comply with the Protocol requirements; and
* Must be willing and able to provide written informed consent at Screening (Visit 1).

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Disease limited to proctitis <15 cm from anal verge;
* Short bowel or malabsorption syndromes;
* Prior intestinal or colon resection surgery (with exception of cholecystectomy or appendectomy);
* Severe/fulminant UC;
* Other forms of inflammatory bowel disease including diagnostic uncertainty by the Investigator, or functional gastrointestinal disorders;
* Positive stool test for parasites, bacterial pathogens, or Clostridium difficile;
* Use of any of the following treatments:

  * Oral 5-ASA products at a dose >3.0 g per day (unless the use is currently stable and anticipated to remain stable during the study);
  * Aspirin or other nonsteroidal anti-inflammatory drugs (except aspirin for cardioprotective reasons at a dose of ≤325 mg per day);
  * Loperamide and other antidiarrheal agents or probiotics;
  * Antibiotics or other antibacterial treatment (unless an ophthalmic or otic antibiotic preparation, or a topical antibiotic for skin infection);
  * Faecal Matter Transplant (FMT) or administration of Vowst®, Rebiotix®, or other Live Biotherapeutic Product (LBP);
  * Intravenous or intramuscular corticosteroids;
  * Oral corticosteroids >10 mg prednisolone or equivalent per day;
  * Any drugs formulated for rectal administration and/or interventions;
  * Immunomodulating or immunosuppressing drugs (unless the use is currently stable and anticipated to remain stable during the study);
  * Biologics, ozanimod, etrasimod, tofacitinib, filgotinib, or upadacitinib; or
  * Proton pump inhibitors (PPIs) or H2 blockers.
* Patients whose disease has not responded to or lost response to 2 or more advanced therapies (biologics or small molecules);
* Significant liver impairment;
* Concurrent primary sclerosing cholangitis;
* Clinically significant hematological function abnormalities;
* Known hypersensitivity, intolerance, or contraindication to oral vancomycin, MB310, and/or any excipients;
* History of, or known malignancy (unless adequately treated (i.e., cured) basal cell carcinoma or squamous cell carcinoma of the skin, or cervical intraepithelial neoplasia or carcinoma in situ of the cervix with no evidence of recurrence within 5 years prior to Screening);
* Any infectious disease (HIV is allowed where certain protocol-specified criteria are met);
* Significant cardiovascular condition;
* Involvement in another clinical study (unless observational) within 4 weeks of Screening from the last dose of study drug or 5 half-lives, whichever is longer; or
* Any other clinically relevant or poorly controlled, unstable condition that would confound study endpoints or adversely affect patient safety or compliance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-09-27 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and causality of adverse events (AEs), treatment-emergent AES, AEs of Scientific Interest and SAEs | From Visit 1 to End of Follow-Up (12 weeks after the last dose of study treatment)
Incidence of treatment-emergent clinically significant changes in laboratory parameters, based on haematology, clinical chemistry, and urinalysis test results | From Visit 1 to End of Follow-Up (12 weeks after the last dose of study treatment)
Incidence of treatment-emergent clinically significant changes in 12-lead ECG parameters, vital signs, and physical examination | From Visit 1 to End of Follow-Up (12 weeks after the last dose of study treatment)

SECONDARY OUTCOMES:
Percentage of patients achieving clinical remission at Day 91 | Day 91
  Clinical remission defined as a Modified Mayo Score (MMS) 0 to 2 with endoscopic subscore of 0 or 1
Percentage of patients achieving steroid-free remission at Day 91 | Day 91
  No steroid exposure at Day 91 with a MMS score of 0 to 2 with endoscopic subscore of 0 or 1
Percentage of patients achieving persistent steroid-free remission at Day 91 | Day 64 to Day 91
  No steroid exposure between Day 64 and Day 91 with a MMS score of 0 to 2 with endoscopic subscore of 0 or 1
Percentage of patients achieving clinical response at Day 91 | Day 91
  Clinical response defined as a decrease in MMS by 2 or more points and at least a 30% reduction from baseline, and a decrease in the rectal bleeding subscore of 1 or more or an absolute rectal bleeding subscore of 0 or 1
Percentage of patients achieving endoscopic improvement at Day 91 | Day 91
  Endoscopic improvement is defined as a decrease in MMS endoscopic subscore by 1 or more point from baseline
Percentage of patients who achieve clinical improvement at Day 64 (Visit 10) and Day 91 (Visit 11) | Day 91
  Clinical improvement defined as a decrease in Partial Mayo Score (pMayo) of 2 or more points from baseline
Time to clinical improvement | End of Follow-Up (12 weeks after the last dose of study treatment)
  Clinical improvement defined as a decrease in Partial Mayo Score (pMayo) of 2 or more points from baseline
Engraftment of MB310 bacteria into patients' intestinal microbial community | Up to End of Follow-Up (12 weeks after the last dose of study treatment)
  Measurement of MB310 strain colonisation in stool samples using a qPCR-based approach.

CONTACTS AND LOCATIONS:
Locations (18):
- Austria (4):
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Klinikum Klagenfurt am Woerthersee, Klagenfurt
  - Uniklinikum Salzburg, Salzburg
  - Medizinische Universitaet Wien, Vienna
- Bulgaria (5):
  - Acibadem City Clinic, Tokuda Hospital, Sofia
  - Diagnostic Consulting Center Convex EOOD, Sofia
  - Medical Center Rusemed EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment, Stara Zagora
  - Diagnostic-Consulting Center, Varna
- Poland (5):
  - Centrum Medyczne Kermed, Bydgoszcz
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - Panstwowy Instytut Medyczny MSWiA - Klinika Gastroenterologi i Chorob Wewnetrznych, Warsaw
  - Warsaw IBD Point, Warsaw
  - Wojskowy Instytut Medyczny - Panstwowy Instytut Badawczy, Klinika Gastroenterologii i Chorob Wewnetrznych, Warsaw
- United Kingdom (4):
  - University Hospital Birmingham, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - St George's Hospital, London
  - Royal Victoria Infirmary, Newcastle